CLINICAL TRIAL: NCT03313128
Title: SaniVac Trial: An Assessment of Oral Rotavirus Vaccine Performance Among Infants Enrolled in a Controlled Before-after Study in Low-income Neighbourhoods of Maputo, Mozambique
Brief Title: SaniVac Trial - Sanitation and Oral Rotavirus Vaccine Performance
Status: Completed | Type: Observational
Sponsor: London School of Hygiene and Tropical Medicine (Other)
Collaborators: Instituto Nacional de Saúde, Mozambique (Other Government); Georgia Institute of Technology (Other); Centers for Disease Control and Prevention (U.S. Federal Agency)
Responsible Party: Sponsor
Other Study IDs: QA919
Record Dates: First submitted 2017-10-06; First posted 2017-10-18 (Actual); Last update posted 2025-12-26 (Actual); Status verified 2025-12

CONDITIONS: Rotavirus Infections; Environmental Enteric Dysfunction; Enteric Infections
MeSH Terms: conditions — Rotavirus Infections | interventions — Sanitation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Historic intervention: Infants born into the historic intervention arm of sanitation trial (NCT02362932)
  Interventions: Other: Sanitation
- Historic control: Infants born into the historic control arm of sanitation trial (NCT02362932)

INTERVENTIONS:
Other: Sanitation — Improved sanitation facility
  Groups: Historic intervention

SUMMARY:
This is a controlled cohort study to assess the effect of improved sanitation on oral rotavirus vaccine performance in low-income urban neighbourhoods of Maputo, Mozambique. The specific hypotheses are that: (1) access to improved sanitation is associated with increased oral rotavirus vaccine immunogenicity; (2) enteric infection concurrent to oral rotavirus vaccination is associated with reduced oral rotavirus vaccine immunogenicity; and (3) Environmental Enteric Dysfunction is associated with reduced oral rotavirus vaccine immunogenicity.

Pregnant women will be enrolled from the intervention and control arms of a previous sanitation trial (NCT02362932) post-intervention and will be enrolled at no later than eight months' gestation and then followed to 4 months of age of the infant. Blood samples and faeces will be taken from the infant at the time of administration of the first dose of the oral rotavirus vaccine and four weeks after the second dose of the vaccine.

The primary outcome of interest in the study is oral rotavirus vaccine immunogenicity among participating vaccinated infants. Seroconversion is defined as a ≥ fourfold rise in serum anti-rotavirus IgA titers between first dose of oral RV vaccine and 4 weeks (+/- 1 week) after second dose of oral RV vaccine. Enteric infections are defined as the presence of ≥ 1 of the following enteric infections in stool: adenovirus 40/41, rotavirus A, norovirus GI/GII, Salmonella spp. (including serovars Typhi and Paratyphi), Campylobacter spp. (C. jejuni, C. coli, C. lari), Shigella spp. (S. boydii, S. sonnei, S. flexneri, S. dysenteriae), Clostridium difficile Toxin A/B, enterotoxigenic Escherichia coli (ETEC) LT/ST, E. coli O157, Shiga-like toxin-producing E. coli (STEC) stx1/stx2, Yersinia enterocolitica, Vibrio cholerae, Giardia lamblia, Entamoeba histolytica, and Cryptosporidium spp. (C. parvum, C. hominis). Environmental Enteric Dysfunction is measured via a combined disease activity score including faecal markers of intestinal inflammation and permeability: neopterin, α-1 antitrypsin, and myeloperoxidase in stool.

ELIGIBILITY:
Inclusion Criteria:

1. Mother residing in an intervention or control compound of a previous sanitation trial (NCT02362932) for at least 6 months prior to recruitment and not intending to switch study compound over the next 9 months
2. Mother being pregnant and having gestational age between 3 and 9 months or being puerperal (up to 40 days postpartum)
3. Mother planning to use the prenatal care, delivery and vaccination services provided by the Ministry of Health of Mozambique
4. Mother able to understand and complete the informed consent process and allow your newborn to participate in the study
5. Mother at least 16 years of age
6. Infant eligible to receive rotavirus vaccination

Exclusion criteria:

1. Infant whose medical team considers that they cannot be part of the study
2. Infant with complications associated with gestation, childbirth or postpartum, including congenital malformations
3. Infant with any medical, psychiatric or social condition, occupational reason, or other responsibility on the part of the pregnant woman, which, in the opinion of the investigator, is a contraindication to protocol compliance or impedes the participant's ability to give informed consent
4. Infant who has already received the rotavirus vaccine

Min Age: 16 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Gender Based: Yes — Pregnant women and their infants
Study Population: Pregnant women of gestational age between 3-9 months (and postpartum) residing in the historic intervention and control compounds of a previous sanitation trial (NCT02362932) and their descendant(s) [infant(s)] of that pregnancy.
Sampling Method: Probability Sample
Enrollment: 261 (Actual)
Dates: Start 2017-10-05 (Actual); Primary Completion 2024-12-12 (Actual); Study Completion 2024-12-12 (Actual)

PRIMARY OUTCOMES:
Oral rotavirus vaccine seroconversion | Approx. 16 weeks age of infant (4 weeks after second dose of oral rotavirus vaccine)
  Seroconversion is defined as a ≥ fourfold rise in serum anti-rotavirus IgA titers between first dose of oral RV vaccine and 4 weeks (+/- 1 week) after second dose of oral RV vaccine

SECONDARY OUTCOMES:
Enteric infection | Approx. 8 weeks age of infant (date of first dose of oral rotavirus vaccine)
  Enteric infections are defined as the presence of ≥ 1 of the following enteric infections in stool: adenovirus 40/41, rotavirus A, norovirus GI/GII, Salmonella spp. (including serovars Typhi and Paratyphi), Campylobacter spp. (C. jejuni, C. coli, C. lari), Shigella spp. (S. boydii, S. sonnei, S. flexneri, S. dysenteriae), Clostridium difficile Toxin A/B, enterotoxigenic Escherichia coli (ETEC) LT/ST, E. coli O157, Shiga-like toxin-producing E. coli (STEC) stx1/stx2, Yersinia enterocolitica, Vibrio cholerae, Giardia lamblia, Entamoeba histolytica, and Cryptosporidium spp. (C. parvum, C. hominis).
Environmental Enteric Dysfunction | Approx. 8 weeks age of infant (date of first dose of oral rotavirus vaccine)
  EED is measured via a combined disease activity score including faecal markers of intestinal inflammation and permeability: neopterin, α-1-antitrypsin, and myeloperoxidase in stool.

CONTACTS AND LOCATIONS:
Overall Officials: Oliver D Cumming, MSc, Principal Investigator — London School of Hygiene and Tropical Medicine; Edna Viegas, MD, Principal Investigator — Centro de Investigação em Saúde da Polana Caniço (CISPOC)
Locations (1):
- Centro de Investigação em Saúde da Polana Caniço (CISPOC), Maputo, Mozambique

IPD SHARING:
Plan to Share IPD: Undecided